CLINICAL TRIAL: NCT03073226
Title: A Prospective Study Comparing the Accuracy of Olympus Lucera Spectrum Technology vs Olympus Lucera Elite Technology in the in Vivo Diagnosis of Barrett's Oesophagus and Colorectal Polyps: The ELITE Study
Acronym: ELITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: PHT/2015/105
Record Dates: First submitted 2017-02-28; First posted 2017-03-08 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Barrett Esophagus; Polyps
MeSH Terms: conditions — Barrett Esophagus; Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Barrett's surveillance Olympus Spectrum (Experimental): Barrett's surveillance with Olympus Spectrum.
  Interventions: Device: Olympus Spectrum
- Barrett's Surveillance Olympus Elite (Experimental): Barrett's surveillance with Olympus ELITE.
  Interventions: Device: Olympus Elite
- Polyp Surveillance Olympus Spectrum (Experimental): Colonic polyp surveillance/screening with Olympus Spectrum.
  Interventions: Device: Olympus Spectrum
- Polyp Surveillancewith Olympus ELITE. (Experimental): Colonic polyp surveillance/screening with Olympus ELITE.
  Interventions: Device: Olympus Elite

INTERVENTIONS:
Device: Olympus Elite — New generation Olympus endoscope
  Arms: Barrett's Surveillance Olympus Elite; Polyp Surveillancewith Olympus ELITE.
Device: Olympus Spectrum — Current generation Olympus endoscope
  Arms: Barrett's surveillance Olympus Spectrum; Polyp Surveillance Olympus Spectrum

SUMMARY:
Barrett's oesophagus is a condition where the lining of the oesophagus (gullet) wall changes. People with Barrett's oesophagus are at risk of developing oesophageal cancer but can have regular checkups to detect changes before they progress to cancer. Every two years patients with Barrett's are offered examination by passing a fibreoptic tube into the oesophagus (gastroscopy) to remove small tissue samples (biopsies), which are examined in the laboratory to check for changes.

Bowel cancer is the third most common cancer in the UK, and the second leading cause of cancer deaths. Prevention and early detection are the most effective strategies of dealing with bowel cancer. Most cancers develop from benign polyps (growths) in the bowel. Polyps are common and have the potential of developing into cancer over the course of many years.

Patients with a prior diagnosis of Barrett's oesophagus and colonic polyps undergo regular endoscopic examinations known as surveillance endoscopies. This is done to detect changes in the cells of Barrett's oesophagus or further polyps. Current practice is to capture recorded videos of Barrett's surveillance examinations and still images of polyps prior to their removal.

Endoscope technology continues to advance. These newly developed technologies are marketed to have claims of superiority in performance over preceding generations often without the back up of scientific data but at a significant financial cost. The aim of this study is to use endoscopic images and videos recorded as part of routine clinical practice to compare the current version of Olympus endoscopes with the new version launched by the company.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending for Barrett's surveillance OR
* Patients attending for colonic polyp surveillance or screening
* Patients are willing and able to give informed consent.

Exclusion Criteria:

* Polyp syndromes (eg FAP or Lynch Syndrome)
* Known history of IBD

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2016-02-06 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-02-06 (Actual)

PRIMARY OUTCOMES:
Sensitivity | Baseline and 1 day
  Difference in the sensitivity of in vivo lesion characterisation between Lucera Elite vs Lucera Spectrum as compared to final histology.

SECONDARY OUTCOMES:
Difference in clarity of images/videos between Lucera Elite and Lucera Spectrum technology. | Baseline and 1 day
  Difference in clarity of images/videos between Lucera Elite and Lucera Spectrum technology.
Sensitivity of Dual Focus technology | Baseline and 1 day
  Difference in sensitivity of lesion characterisation when using dual focus technology.
Endoscopists confidence | Baseline and 1 day
  Difference in endoscopists' confidence scores in lesion characterisation between new and current technologies.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Alexandra Hospital, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No current plan